CLINICAL TRIAL: NCT02833558
Title: Randomised Controlled Trial Comparing Purastat® to Standard Therapy for Haemostasis Control During Endoscopic Submucosal Dissection
Brief Title: Purastat® vs Standard Therapy for Haemostasis During Endoscopic Submucosal Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHT/2015/106
Record Dates: First submitted 2016-06-29; First posted 2016-07-14 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Gastrointestinal Haemorrhage
Keywords: Endoscopy, Gastrointestinal; Endoscopic Submucosal Dissection; Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hemorrhage | interventions — Electrocoagulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PuraStat® (Experimental): Interventional arm: PuraStat® applied through a catheter delivery system via the endoscope is used to stop bleeding during ESD.
  Interventions: Device: PuraStat®
- Standard Electrocautery (Other): Control arm where standard electrocautery delivered via the endoscopic knife tip or coag grasper is used to achieve haemostasis during ESD
  Interventions: Procedure: Electrocautery

INTERVENTIONS:
Device: PuraStat® — PuraStat® gel is applied through a safe catheter delivery system (via endoscope) over the bleeding point
  Arms: PuraStat®
Procedure: Electrocautery — Electrocautery (coagulation current) to stop bleeding during ESD
  Arms: Standard Electrocautery

SUMMARY:
Endoscopic submucosal dissection (ESD) is an endoscopic resection technique used to treat superficial neoplasia in the gastrointestinal tract. Bleeding is a commonly encountered problem during submucosal dissection and is usually managed with electrocautery. However, this does carry a risk of deep thermal injury and perforation.

PuraStat® is a novel extracellular scaffold matrix of amino acids that forms a transparent adherent barrier when applied to a bleeding point.

The aim of this trial is to study the use of PuraStat® in reducing the need for thermal haemostasis during ESD.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is an endoscopic technique that involves the use of an endoscopic knife to gently peel off a superficial neoplasia of any size in an en-bloc fashion. It meets the principles of onco-surgery and is associated with excellent outcomes. A difficulty however with the technique is control of bleeding during the procedure. The GI mucosa is a vascular territory and the current method of managing intraprocedural bleeding is electrocautery using either the endoscopic knife itself or the coag grasper. This introduces a thermal injury to the bowel wall and carries the risk of causing a perforation or causing pain. Furthermore, it requires precise targeting of the bleeding vessel. Practically this can be challenging, particularly if the coag grasper is needed which is a bulky device and can be difficult to apply precisely in some locations.

PuraStat® (3-D Matrix Ltd, Tokyo) is a liquid which is applied to a bleeding area which acts rapidly to form a gel coat which induces haemostasis. This transparent adherent barrier permits further endoscopic therapy to be performed. It can be applied in the general area of bleeding and does not require precise application to the exact point of bleeding. It is applied through a small catheter placed through the biopsy channel of the endoscope which can be used in very small spaces.

PuraStat® is licensed as a CE marked device for use in exudative haemorrhage from vessels in solid organs and within the GI tract. Given this indication, the role of PuraStat in ESD needs to be explored as it could reduce the need for thermal haemostasis. This would be of significant clinical benefit during ESD.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above.
* An ESD is attempted for clinical indications approved by MDT.
* Oesophageal or colonic lesion 2-5cm in size
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Known coagulopathy likely to affect risk of bleeding
* Submucosal tumour
* Anticoagulation or anti-platelet therapy (apart from single modality aspirin or clopidogrel) which cannot be stopped for clinical reasons
* Patient preference

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
The number of times intraprocedural heat therapy is used to achieve haemostasis in ESD in both the PuraStat® and control arms of the study | Measured during the ESD procedure

SECONDARY OUTCOMES:
The length of the procedure in the PuraStat® and control arm of the study | Measured during the ESD procedure
The number of patients with delayed bleeding (bleeding within 28 days) in both the PuraStat® and control arm of the study | 28 days
Wound healing in the PuraStat® and control arm at 6 weeks post ESD | 6 weeks
  Wound healing will be measured at endoscopy using qualitative descriptor categories (active ulceration, healing ulceration, scarring or complete mucosal healing). There is no standard definition to qualify ulcer healing post ESD but these categories have previously been used by Uraoka et al in a similar study published in Gastrointestinal Endoscopy (Vol 83, No 6:2016.1259-1264).
Number of adverse events in the PuraStat® and control arm of the study | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhandari, MBBS, MD, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmputh Hospitals NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes